CLINICAL TRIAL: NCT03232294
Title: Effect of Fetal Front-abdominal Wall Thickness on Birth Weight and Perinatal Outcome at 24-26. Gestational Weeks
Brief Title: Fetal Front-abdominal Wall Thickness and Perinatal Outcome
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf MADENDAG, principal investigator, Kayseri Education and Research Hospital
Other Study IDs: 2017/222
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Fetal Macrosomia; Abdominal Wall Mass; Perinatal Problems
Keywords: fetal macrosomia; fetal abdominal wall thickness; subcutaneous adipose tissue
MeSH Terms: conditions — Fetal Macrosomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the study group: A total of 96 women with low risk pregnancy coming to the clinic for a routine antenatal examination in 26-28th gestational weeks were included to this study

SUMMARY:
Abnormal fetal development such as macrosomia can cause some complications on both fetus and mother.The measurement of fetal anterior abdominal wall thickness (FAWT) is an easy examination that it can be obtained during an examination of a pregnant woman by ultrasound. Macrosomia for fetus can lead to some morbidities. It can affect perinatal outcome and increase childbirth complications and operative birth. There are some studies scrutinizing the relationship between FAWT and diabetes in the literature. However there are few studies which scrutinize effect of FAWT on both abnormal fetal development and adverse perinatal outcomes in non-diabetic pregnancies and non high risk pregnancies. Hence the investigators wonder if FAWT can anticipate birth-weight or macrosomic infant or perinatal outcome regarding with macrosomia in the second trimester.

ELIGIBILITY:
Inclusion Criteria:

A total of 96 women with low risk pregnancy coming to our clinic for a routine antenatal examination in 26-28th gestational weeks were included to this study and performed 75 gr- oral glucose tolerance test (OGTT).

Exclusion Criteria:

The participants with a positive 75-g OGTT were excluded. Additionally those following criteria were accepted as the exclusion criteria of this study: hypertension, preeclampsia, diabetes, fetal distress, fetal anomaly, multiple pregnancy, preterm labor, preterm premature rupture of membrane, placenta previa, polyhydramnios and intrauterine fetal growth restriction.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 96 women with low risk pregnancy coming to our clinic for a routine antenatal examination in 26-28th gestational weeks were included to this study
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
The relationship between fetal abdominal wall thickness and macrosomia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: YUSUF MADENDAG, Principal Investigator — Kayseri Education and Research Hospital